CLINICAL TRIAL: NCT06853574
Title: Changes in Ventriculo-arterial Coupling and Myocardial Work During Treatment of Sepsis and Septic Shock: a Prospective Interventional Study
Brief Title: Ventriculo-arterial Coupling and Myocardial Work in Sepsis and Septic Shock
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General and Teaching Hospital Celje (Other)
Responsible Party: Principal Investigator, Matej Podbregar, Prof. Dr. Matej Podbregar, General and Teaching Hospital Celje
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 70/2025/6-1
Record Dates: First submitted 2025-01-31; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; myocardial work; ventriculo-arterial coupling; ICU; intensive care
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluids (Active Comparator): The patients will be included in this arm on admission basing on the absence of peripheral edema, presence of apical A lines at lung ultrasound, inferior vena cava width < 2 cm and velocity-time integral (VTI) variation > 10%.
  If the fluid therapy will not be effective, patients will also receive vasopressors.
  Interventions: Drug: Fluid therapy; Drug: Noradrenaline infusion
- No fluids (Active Comparator): The patients will be included in this arm on admission basing on the presence of peripheral edema, presence of apical B lines at lung ultrasound, inferior vena cava width > 2 cm and velocity-time integral (VTI) variation < 10%.
  In this arm the patients will receive vasopressors with an initial mean arterial pressure target of 65 mmHg; then the investigators will target to 80-85 mmHg to observe tha changes in ventriculo-arterial coupling.
  Interventions: Drug: Noradrenaline infusion

INTERVENTIONS:
Drug: Fluid therapy — Infusion of 8 ml/Kg/30' or 16 ml/kg/60' of fluids.
  Arms: Fluids
Drug: Noradrenaline infusion — dosage will be titrated in order to obtain mean arterial pressure target
  Other Names: Vasopressin infusion

SUMMARY:
Sepsis is a term which describes an excessive response of the body to an infection and, if not promptly treated, can turn into septic shock a condition in which the organs don't receive enough oxygen to satisfy their needs. The aim of the study is to assess how the treatment of sepsis and septic shock will modify myocardial work and ventriculo-arterial coupling, that can be considered as indicators of ventricular and arterial performance efficacy respectively. Each patient will be treated according to updated guidelines for sepsis and septic shock management, they will voluntarily be enrolled and they can decide to withdraw in each moment without any consequence on their treatment. The investigators, after receiving the consent, will collect patients' data, take blood samples and perform ultrasound measurements and then will start the treatment which can be based on fluids infusion, vasopressors or both. The investigators think that a modern cardiovascular assessment approach can be used to individually set the optimal blood pressure target in sepsis and septic shock with the combined evaluation of myocardial work and ventriculo-arterial coupling.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* sepsis
* septic shock

Exclusion Criteria:

* lack of consent
* less than 18 years old
* pregnancy
* more than moderate aortic stenosis ( aortic valve area (AVA) < 1.4 cm2, aortic valve area indexed (AVAi) < 0.85, doppler velocity index (DVI) < 0.5)
* more than mild mitral regurgitation (vena contracta (VC) width <= 3 mm, mitral regurgitation (MR) effective regurgitant orifice area (EROA) < 20, MR regurgitant volume (RegV) < 30 ml)
* cardiac arrythmias (e.g. atrial fibrillation/flutter, frequent ventricular and supraventricular or nodal activity)
* renal replacement therapy
* other than continous modes of mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Changes in ventriculo-arterial coupling | From enrollment to 24 hours after treatment start
  ventricular coupling will be analyzed on admission and its changes after treatment will be observed. To analyze ventriculo-arterial coupling, invasive blood pressure through either a radial or femoral arterial line will be collected and then data will be plotted into iElastance app available on smartphones to get the also knows as single beat determination ventriculo-arterial coupling.
Changes in myocardial work | From enrollment to 24 hours after treatment start
  Myocardial work will be analyzed on admission and its changes after treatment will be observed. To realize this, a transthoracic cardiac ultrasound will be performed and the images will be transferred to EchoPAC from General Electrics (GE) to get the pressure-volume strain analysis also known as myocardial work.

SECONDARY OUTCOMES:
Mean arterial pressure optimal target | From enrollment to 24 hours after treatment start
  The study aims to identify the optimal mean arterial pressure (MAP) target in sepsis and septic shock with the combined evaluation of myocardial work and ventriculo-arterial coupling. To realize this, invasive blood pressure through either a radial or femoral arterial line will be collected and then data will be plotted into iElastance app available on smartphones to get the also knows as single beat determination ventriculo-arterial coupling.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Celje, Celje, Slovenia

IPD SHARING:
Plan to Share IPD: No
Only the investigators involved in the study at General Hospital in Celje - Internal Intensive Care Unit (SBC - OIIM) will manage participant data.

REFERENCES:
- [Background] Sunagawa K, Sagawa K, Maughan WL. Ventricular interaction with the loading system. Ann Biomed Eng. 1984;12(2):163-89. doi: 10.1007/BF02584229. PMID 6507965
- [Background] Kakihana Y, Nishida O, Taniguchi T, Okajima M, Morimatsu H, Ogura H, Yamada Y, Nagano T, Morishima E, Matsuda N; J-Land 3S Study Group. Efficacy and safety of landiolol, an ultra-short-acting beta1-selective antagonist, for treatment of sepsis-related tachyarrhythmia (J-Land 3S): a multicentre, open-label, randomised controlled trial. Lancet Respir Med. 2020 Sep;8(9):863-872. doi: 10.1016/S2213-2600(20)30037-0. Epub 2020 Mar 31. PMID 32243865
- [Background] Morelli A, Ertmer C, Westphal M, Rehberg S, Kampmeier T, Ligges S, Orecchioni A, D'Egidio A, D'Ippoliti F, Raffone C, Venditti M, Guarracino F, Girardis M, Tritapepe L, Pietropaoli P, Mebazaa A, Singer M. Effect of heart rate control with esmolol on hemodynamic and clinical outcomes in patients with septic shock: a randomized clinical trial. JAMA. 2013 Oct 23;310(16):1683-91. doi: 10.1001/jama.2013.278477. PMID 24108526
- [Background] Nasrollahi-Shirazi S, Sucic S, Yang Q, Freissmuth M, Nanoff C. Comparison of the beta-Adrenergic Receptor Antagonists Landiolol and Esmolol: Receptor Selectivity, Partial Agonism, and Pharmacochaperoning Actions. J Pharmacol Exp Ther. 2016 Oct;359(1):73-81. doi: 10.1124/jpet.116.232884. Epub 2016 Jul 22. PMID 27451411
- [Background] Zhou X, Pan J, Wang Y, Wang H, Xu Z, Zhuo W. Left ventricular-arterial coupling as a predictor of stroke volume response to norepinephrine in septic shock - a prospective cohort study. BMC Anesthesiol. 2021 Feb 17;21(1):56. doi: 10.1186/s12871-021-01276-y. PMID 33596822
- [Background] Chen CH, Fetics B, Nevo E, Rochitte CE, Chiou KR, Ding PA, Kawaguchi M, Kass DA. Noninvasive single-beat determination of left ventricular end-systolic elastance in humans. J Am Coll Cardiol. 2001 Dec;38(7):2028-34. doi: 10.1016/s0735-1097(01)01651-5. PMID 11738311
- [Background] Zhou X, Zhang Y, Pan J, Wang Y, Wang H, Xu Z, Chen B, Hu C. Optimizing left ventricular-arterial coupling during the initial resuscitation in septic shock - a pilot prospective randomized study. BMC Anesthesiol. 2022 Jan 21;22(1):31. doi: 10.1186/s12871-021-01553-w. PMID 35062874
- [Background] Antonini-Canterin F, Poli S, Vriz O, Pavan D, Bello VD, Nicolosi GL. The Ventricular-Arterial Coupling: From Basic Pathophysiology to Clinical Application in the Echocardiography Laboratory. J Cardiovasc Echogr. 2013 Oct-Dec;23(4):91-95. doi: 10.4103/2211-4122.127408. PMID 28465893
- [Background] Andrei S, Bahr PA, Berthoud V, Popescu BA, Nguyen M, Bouhemad B, Guinot PG. Diuretics depletion improves cardiac output and ventriculo-arterial coupling in congestive ICU patients during hemodynamic de-escalation. J Clin Monit Comput. 2023 Aug;37(4):1035-1043. doi: 10.1007/s10877-023-01011-7. Epub 2023 Apr 25. PMID 37097337
- [Background] Bischoff AR, Stanford AH, McNamara PJ. Short-term ventriculo-arterial coupling and myocardial work efficiency in preterm infants undergoing percutaneous patent ductus arteriosus closure. Physiol Rep. 2021 Nov;9(22):e15108. doi: 10.14814/phy2.15108. PMID 34806325
- [Background] Demailly Z, Besnier E, Tamion F, Lesur O. Ventriculo-arterial (un)coupling in septic shock: Impact of current and upcoming hemodynamic drugs. Front Cardiovasc Med. 2023 May 30;10:1172703. doi: 10.3389/fcvm.2023.1172703. eCollection 2023. PMID 37324631
- [Background] Rehn M, Chew MS, Olkkola KT, Ingi Sigurethsson M, Yli-Hankala A, Hylander Moller M. Surviving sepsis campaign: International guidelines for management of sepsis and septic shock in adults 2021 - endorsement by the Scandinavian society of anaesthesiology and intensive care medicine. Acta Anaesthesiol Scand. 2022 May;66(5):634-635. doi: 10.1111/aas.14045. Epub 2022 Mar 6. PMID 35170043

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT06853574/Prot_SAP_ICF_000.pdf